CLINICAL TRIAL: NCT02592564
Title: The Brain´s Plasticity and Change in Cellular Aging After Internet-delivered Cognitive Behavior Therapy for Social Anxiety Disorder
Brief Title: Brain Plasticity and Cellular Aging After Internet-delivered CBT for Social Anxiety Disorder
Acronym: UMEII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Umeå University (Other); Uppsala University (Other); Stockholm University (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristoffer NT Månsson, PhD, Stockholm University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMESTUDIEN-II
Record Dates: First submitted 2015-10-23; First posted 2015-10-30 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Anxiety Disorders; Social Anxiety Disorder
Keywords: Magnetic Resonance Imaging; Cognitive Behavior Therapy; Telomerase; Telomere Length, Mean Leukocyte
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychological treatment (Experimental): Psychological treatment during 9 weeks.
  Interventions: Behavioral: Internet-delivered cognitive behavior therapy

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavior therapy — Internet-delivered cognitive behavior therapy for social anxiety disorder. Similar to previous studies in our research group, the treatment will be delivered during 9 weeks. Each week the participant will be introduced to a module containing text material and homework assignments. The participants will receive feedback via text by a clinical psychologist once a week.
  Other Names: Internet-delivered CBT

SUMMARY:
This study evaluates underlying psychological and biological mediators in Internet-delivered cognitive behavior therapy for adults with social anxiety disorder.

DETAILED DESCRIPTION:
Internet-delivered cognitive behavior therapy for social anxiety disorder has previously demonstrated to target and affect the brain´s fear network, typically neural response in the amygdala ameliorate after effective psychological treatment. Commonly, neuroimaging studies have performed brain imaging at pre- and post-intervention, yet, longitudinal study designs including several repeated measures of neural response over the course of treatment are currently missing in anxiety disorder. In the current study the participants will undergo magnetic resonance imaging (MRI) at four occasion. a) Twice before treatment initiation (9 weeks apart), b) at week 4 (during treatment), c) and directly after treatment termination.

Biological aging can be quantified at the individual cell level by measuring telomere length in peripheral immune cells (leukocytes). Telomeres are located at the end of each chromosome and protect the genetic material during cell division. Telomerase is an enzyme that can lengthen telomeres, and have in this way a protective function against accelerated cellular aging. Variations in these bodily processes have been associated with psychiatric manifestations such as anxiety and depression. In the current study the participant´s telomere length and telomerase activity will be assessed at three occasion. a) Twice before treatment initiation (9 weeks apart), and b) directly after treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* Social Anxiety Disorder as primary diagnosis (DSM-5)
* Otherwise somatically healthy
* Willingness to participate in a symptom provocation brain imaging trial

Exclusion Criteria:

* Concurrent psychological treatment
* Treatment of social anxiety within the three months preceding the study
* Chronic use of prescribed medication that could influence the results (anxiolytic or antidepressant drugs, certain hypnotics or herbs like St Johns Wort)
* Contraindications for MRI investigation (implants or other metal objects in the body, brain and heart operations)
* Pregnancy or planned pregnancy during the first 6 months of the study period
* Postmenopausal women
* Any neurological disorders
* Depressive symptoms, as determined by scoring more than 20 on the MADRS questionnaire (self-report version)
* Suicidal ideation (scoring more than 2) on the self-report version of MADRS, item 9
* Suicide at moderate risk (MINI v7)
* Bipolar disorder (MINI v7)
* Psychotic syndromes (MINI v7)
* Substance abuse disorders (MINI v7)
* Alcohol abuse (MINI v7)
* Any eating disorder (MINI v7)
* Antisocial personality disorder (MINI v7)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Clinically Global Impression-Improvement scale (CGI-I; Change from baseline) | At week 20 (post-treatment), and at 6, 12, and 60 months
  Clinician administrated telephone-interview to determine the participant´s treatment response rates (very much worse to very much improved)
Liebowitz Social Anxiety Scale, Self-report version (LSAS-SR; Change from baseline) | Screening, Baseline 1 (week 0), Baseline 2 (week 9), weekly during treatment (week 10-19), week 20 (post-treatment), and at 6, 12, and 60 months
  Self reported social anxiety symptoms on fear (scoring 0-3) and avoidance (scoring 0-3) in 24 social situations.

SECONDARY OUTCOMES:
Clinically Global Impression-Severity scale (CGI-S) | Screening, week 20 (post-treatment), and at 6, 12, and 60 months
  Clinician administrated telephone-interview to determine the participant´s severity of illness
Social Phobia Screening Questionnaire (SPSQ) | Screening, week 20 (post-treatment), and at 6, 12, and 60 months
  Self reported social anxiety symptoms on distress (scoring 0-4) in 24 social situations.
Beck Anxiety Inventory (BAI) | Screening, week 20 (post-treatment), and at 6, 12, and 60 months
  Self reported anxiety symptoms
Social Interaction Anxiety Scale (SIAS) | Screening, week 20 (post-treatment), and at 6, 12, and 60 months
  Self reported social anxiety symptoms on distress (scoring 0-4) in 21 social situations.
Social Phobia Scale (SPS) | Screening, week 20 (post-treatment), and at 6, 12, and 60 months
  Self reported social anxiety symptoms on distress (scoring 0-4) in 20 social situations.
Montgomery Åsberg Depression Rating Scale, Self-report version (MADRS-S) | Screening, Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment), and at 6, 12, and 60 months
  Self reported depressive symptoms (scoring 0-6).
Subjective unit of discomfort on fear and distress (SUD) | Before experimental tasks while undergoing MRI, at Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
  Self reported scoring 0-100 on fear and distress separately
Social Probability/Cost Questionnaire | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment), and at 6, 12, and 60 months
  40 items scoring 0 to 8. Foa et al., 1996, J Abnormal Psychology
Quality of Life (QOLI) | Screening, week 20 (post-treatment), and at 6, 12, and 60 months
Social Network Index (SNI) | Baseline 1 (week 0)
  Bickart et al., 2010, Nat Neurosci
Brown Attention-Deficit Disorder Scales (Brown ADD) | Baseline 1 (week 0)
Difficulties in Emotion Regulation Scale (DERS) | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment), and at 6, 12, and 60 months
Treatment Credibility Scale (TCS) | Baseline 2 (week 9), week 13 during treatment
Revised NEO Personality Inventory (NEO-PI-R) | Baseline 1 (week 0)
Insomnia Severity Index (ISI) | Baseline 1 (week 0)
Karolinska Sleep Questionnaire (KSQ) | Baseline 1 (week 0)
State-Trait Anxiety Inventory (STAI-T) | Baseline 1 (week 0)
State-Trait Anxiety Inventory (STAI-S) | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
MINI International Neuropsychiatric Interview | Screening
  Swedish version 7.0.0

OTHER OUTCOMES:
Resting-state fMRI 6 minutes | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
  Salami et al., 2014, PNAS
Self-referential criticism | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
  Blair et al., 2008, Arch Gen Psych
Hariri´s Hammer (emotional face perception) | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
  Hariri et al., 2002, Science
Brain habituation during face perception | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
  Fischer et al., 2003, Brain Research Bulletin
Diffusion Tensor Imaging (DTI) | Baseline 1 (week 0), Baseline 2 (week 9), week 13 during treatment, week 20 (post-treatment)
  Salami et al., 2012, Biochim Biophys Acta
Leukocyte telomere length | Baseline 1 (week 0), Baseline 2 (week 9), week 20 (post-treatment)
  Lindqvist et al., 2015, Neurosci Biobehav Rev
Telomere terminal transferase (telomerase) | Baseline 1 (week 0), Baseline 2 (week 9), week 20 (post-treatment)
  Wolkowitz et al., 2012, Mol Psychiatry

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer NT Månsson, PhD, Principal Investigator — Stockholm University, Karolinska Institutet
Locations (1):
- Umeå university, Umeå, Sweden

REFERENCES:
- [Background] Mansson KN, Carlbring P, Frick A, Engman J, Olsson CJ, Bodlund O, Furmark T, Andersson G. Altered neural correlates of affective processing after internet-delivered cognitive behavior therapy for social anxiety disorder. Psychiatry Res. 2013 Dec 30;214(3):229-37. doi: 10.1016/j.pscychresns.2013.08.012. Epub 2013 Sep 21. PMID 24064198
- [Background] Mansson KN, Frick A, Boraxbekk CJ, Marquand AF, Williams SC, Carlbring P, Andersson G, Furmark T. Predicting long-term outcome of Internet-delivered cognitive behavior therapy for social anxiety disorder using fMRI and support vector machine learning. Transl Psychiatry. 2015 Mar 17;5(3):e530. doi: 10.1038/tp.2015.22. PMID 25781229
- [Background] Lindqvist D, Epel ES, Mellon SH, Penninx BW, Revesz D, Verhoeven JE, Reus VI, Lin J, Mahan L, Hough CM, Rosser R, Bersani FS, Blackburn EH, Wolkowitz OM. Psychiatric disorders and leukocyte telomere length: Underlying mechanisms linking mental illness with cellular aging. Neurosci Biobehav Rev. 2015 Aug;55:333-64. doi: 10.1016/j.neubiorev.2015.05.007. Epub 2015 May 18. PMID 25999120
- [Background] Furmark T, Tillfors M, Marteinsdottir I, Fischer H, Pissiota A, Langstrom B, Fredrikson M. Common changes in cerebral blood flow in patients with social phobia treated with citalopram or cognitive-behavioral therapy. Arch Gen Psychiatry. 2002 May;59(5):425-33. doi: 10.1001/archpsyc.59.5.425. PMID 11982446